CLINICAL TRIAL: NCT01770106
Title: Comparison of the Effect of Denosumab and Alendronate on Bone Density and Microarchitecture in Rheumatoid Arthritis Females With Low Bone Mass: A Randomized Controlled Trial
Brief Title: RA Denosumab on Bone Microstructure Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA-2011.510
Record Dates: First submitted 2013-01-03; First posted 2013-01-17 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Bone density; Bone microarchitecture; HR-pQCT
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Denosumab; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Experimental): Patients in this arm will receive subcutaneous injection of denosumab 60mg every 6 months (1 dose for the study period).
  Interventions: Drug: Denosumab
- Standard treatment (Active Comparator): Patients (n=20) in this arm will receive oral alendronate (Fosamax®)70mg once.
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injection of denosumab 60mg every 6 months (1 dose for study period)
  Other Names: Prolia®
  Arms: Denosumab
Drug: Alendronate — Alendronate 70mg once weekly
  Other Names: Fosamax®
  Arms: Standard treatment

SUMMARY:
The aim of this study is to compare the effects of denosumab and a current standard treatment on cortical and trabecular microarchitecture at the radius and second metacarpal in rheumatoid arthritis (RA) patients with low bone mineral density using high resolution peripheral quantitative computed tomography (HR-pQCT) during a 6-month open-label randomized controlled study. Forty ambulatory Chinese females, who consent to receive alendronate as standard treatment subjective to the randomization, will be enrolled in this study. Subjects will be randomized to 2 arms receiving: 1) subcutaneous injection of denosumab 60mg (Prolia®) every 6 months (n=20), or 2) oral alendronate weekly (Fosamax® once weekly 70 mg, n=20). In addition, all patients will be given a daily calcium supplement (1500mg caltrate /day) and 1 multivitamin tablet per day. Efficacy and safety assessment will be performed at baseline, month 3 and month 6. aBMD of lumbar spine, total hip and non-dominant distal radius will be measured using dual-energy X-ray absorptiometry (DXA) and microarchitecture of bone is measured at the non-dominant distal radius and the second metacarpal bone of the non-dominant hand using HR-pQCT.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, systemic inflammatory disease most typical in women. Generalized osteoporosis is common in RA, at axial and appendicular skeleton and in females and males. Denosumab is a fully humanized IgG monoclonal antibody that targets the receptor activator of nuclear factor κB ligand (RANKL). Denosumab prevents the binding and activation of the RANK receptors on the osteoclasts and hence inhibits osteoclasts formation, activation, function and survival. Denosumab results in more rapid and greater reductions in bone remodeling and correspondingly greater increases in areal bone mineral density (aBMD) at all skeletal sites. Denosumab was approved by FDA in June 2010 for the treatment of postmenopausal women with osteoporosis at high risk of fracture. Denosumab (Prolia®) is also licensed in Hong Kong.

A high-resolution peripheral quantitative computed tomography (HR-pQCT) capable of achieving an isotropic voxel size of 80μm at tolerable radiation doses (3μSv) is available for the assessment of trabecular and cortical microarchitecture at the distal radius and tibia. This technique bears excellent precision for both density and microstructure measures. Denosumab's greater potency in suppressing bone remodeling and greater effect on areal BMD than alendronate, particularly at predominantly cortical sites such as the distal third of the radius, may reflect the differing mechanism of action of these drugs, which, in turn, influence bone microarchitecture.

The aim of this study is to compare the effects of denosumab and a current standard treatment on cortical and trabecular microarchitecture at the radius and second metacarpal in RA patients with low bone mineral density using HR-pQCT during a 6-month open-label randomized controlled study. One bisphosphonate, namely alendronate sodium (or alendronate) is chosen to generate a heterogeneous and comparable active control group. This is a 6-month open-label randomized controlled clinical trial. Forty ambulatory Chinese females, who consent to receive alendronate as standard treatment subjective to the randomization, will be enrolled from the rheumatology clinic of the Prince of Wales Hospital in this study. Subjects will be randomized to 2 groups receiving: 1) subcutaneous injection of denosumab 60mg (Prolia®) every 6 months (n=20), or 2) a standard treatment: oral alendronate weekly (Fosamax® once weekly 70 mg, n=20). In addition, all patients will be given a daily calcium supplement (1500mg caltrate /day) and 1 multivitamin tablet per day. Efficacy and safety assessment will be performed at baseline, month 3 and month 6. aBMD of lumbar spine, total hip and non-dominant distal radius will be measured using dual-energy X-ray absorptiometry (DXA) and microarchitecture of bone is measured at the non-dominant distal radius and the second metacarpal bone of the non-dominant hand using HR-pQCT.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of RA according to the 2010 new 2010 American College of Rheumatology/ European League Against Rheumatism classification criteria
* at an age over 18 years old
* have a lumbar spine, or total hip or distal radius T-score lower than -1.5 by DXA
* without severe deformity in metacarpophalangeal (MCP) joints which would influence the longitudinal assessment of HR-pQCT
* consent to receive alendronate if randomized to standard treatment group.

Exclusion Criteria:

* they have previous use of denosumab, teriparatide, alendronate or other anti-resorptive agents;
* they have a history of recent major gastrointestinal (GI) tract disease (e.g. oesophagitis or GI ulceration) or have experienced any previous adverse reaction to bisphosphonate therapy;
* they are receiving other bone-active drugs, such as hormonal replacement therapy, thyroxine, thiazide and diuretics;
* they have conditions affecting bone metabolism; contraindications to alendronate and denosumab (uncorrected hypocalcemia);
* they have unexplained hypocalcemia;
* they have severe renal impairment or serum creatinine level of >200umol/L;
* they are pregnant or breastfeeding;
* they do not understand Chinese or are incompetent in giving consent.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in bone volumetric density at distal radius at 6th month | Baseline to 6th month
  Bone volumetric density is characterized by average volumetric bone mineral density (BMD) at distal radius by HR-pQCT

SECONDARY OUTCOMES:
Changes from baseline in trabecular bone microarchitecture at distal radius at 6th month | Baseline to 6th month
  Trabecular bone microarchitecture is characterized by trabecular bone volume fraction (BV/TV) at distal radius by HR-pQCT
Changes from baseline in bone volumetric density at the 2nd metacarpal bone at 6th month | Baseline to 6th month
  Volumetric bone density is characterized by average volumetric bone mineral density at the 2nd metacarpal bone measured by HR-pQCT
Changes from baseline in trabecular bone microarchitecture at 2nd metacarpal bone at 6th month | Baseline to 6th month
  Trabecular bone microarchitecture is characterized by trabecular bone volume fraction (BV/TV) at 2nd metacarpal head by HR-pQCT
Changes from baseline in areal bone density at total hip at 6th month | Baseline to 6th months
  Areal bone density at total hip is characterized by areal bone mineral density by DXA.
Changes from baseline in areal bone density at lumbar spine at 6th month | Baseline to 6th month
  Areal bone density at lumbar spine is characterized by areal bone mineral denstiy at lumbar spine by DXA
Changes in areal bone density at distal radius at 6th month | Baseline to 6th month
  Areal bone density is characterized by areal bone mineral density at distal radius by DXA
Changes from baseline in bone volumetric density at distal radius at 3rd month | Baseline to 3rd month
  Bone volumetric density is characterized by average volumetric bone mineral density (BMD) at distal radius by HR-pQCT
Changes from baseline in trabecular bone microarchitecture at distal radius at 3rd month | Baseline to 3rd month
  Trabecular bone microarchitecture is characterized by trabecular bone volume fraction (BV/TV) at distal radius by HR-pQCT
Changes from baseline in bone volumetric density at the 2nd metacarpal bone at 3rd month | Baseline to 3rd month
  Volumetric bone density is characterized by average volumetric bone mineral density at the 2nd metacarpal bone measured by HR-pQCT
Changes from baseline in trabecular bone microarchitecture at 2nd metacarpal bone at 3rd month | Baseline to 3rd month
  Trabecular bone microarchitecture is characterized by trabecular bone volume fraction (BV/TV) at 2nd metacarpal head by HR-pQCT
Changes from baseline in areal bone density at total hip at 3rd month | Baseline to 3rd month
  Areal bone density at total hip is characterized by areal bone mineral density by DXA.
Changes from baseline in areal bone density at lumbar spine at 3rd month | Baseline to 3rd month
  Areal bone density at lumbar spine is characterized by areal bone mineral denstiy at lumbar spine by DXA
Changes in areal bone density at distal radius at 3rd month | Baseline to 3rd month
  Areal bone density is characterized by areal bone mineral density at distal radius by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Lai-Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, N.t., Hong Kong

REFERENCES:
- [Derived] Yue J, Griffith JF, Xiao F, Shi L, Wang D, Shen J, Wong P, Li EK, Li M, Li TK, Zhu TY, Hung VW, Qin L, Tam LS. Repair of Bone Erosion in Rheumatoid Arthritis by Denosumab: A High-Resolution Peripheral Quantitative Computed Tomography Study. Arthritis Care Res (Hoboken). 2017 Aug;69(8):1156-1163. doi: 10.1002/acr.23133. Epub 2017 Jul 10. PMID 27768831